CLINICAL TRIAL: NCT07364084
Title: Self-modulation of the mPFC Using Rt-fMRI NF Training to Improve Negative Anticipation for Future Events
Brief Title: Real-time Neurofeedback Training of the Medial Prefrontal Cortex Based on Imagined Social Support
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Benjamin Becker, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: BAM_lab_NF_06
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Healthy; Neurofeedback
Keywords: real-time neurofeedback; social support; mPFC

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurofeedback training (Experimental): Participants in the neurofeedback training group are instructed to regulate their medial prefrontal cortex activity based on the visual intermittent neurofeedback.
  Interventions: Procedure: real-time fMRI sham-controlled neurofeedback training procedure
- Sham control (Sham Comparator): Participants in the sham control group receive the same instruction and perform the same regulation strategy based on neurofeedback from an unrelated region (i.e. primary motor cortex) which is not involved in episodic imagination in related to social support (a controlled sham region).
  Interventions: Procedure: real-time fMRI sham-controlled neurofeedback training procedure

INTERVENTIONS:
Procedure: real-time fMRI sham-controlled neurofeedback training procedure — real-time fMRI neurofeedback training procedure running on the Turbo Brain voyager (TBV) 4.2 software (Brain Innovation, Maastricht, The Netherlands)

SUMMARY:
Randomized active-sham controlled between-subject real-time fMRI neurofeedback trial aiming to modulate activity in the medial prefrontal cortex (mPFC) to improve subjective negative anticipation.

DETAILED DESCRIPTION:
A double-blinded, placebo-controlled, between-subject design will be employed in this study. In a randomized order, a total of 60 healthy subjects will be recruited and assigned to the experimental group (EG; N=30), which receives real feedback from the medial prefrontal cortex (mPFC), or the sham control group (CG; N=30) which receives sham feedback from an unrelated brain region. Neurofeedback training consists of 1 baseline session without feedback (also as a localizer task), 4 training sessions with intermittent feedback and 1 transfer session without feedback. Each NF run includes 5 regulation blocks and 5 baseline blocks. Each trial starts with a jittered fixation cross (2~8 s), a modulation block (i.e. regulation or baseline; 30 s) without continous feedback, and a intermittent feedback period (4s) to display the mean activiation of the mPFC/control region during the regulation block compared with baseline block. Objectives are to determine (1) if subjects in the neurofeedback (NF) group can gain volitional control over the mPFC activation using imagined social support as regulation strategy, (2) whether successful increased modulation of the mPFC could improve negative anticipation and sense of control for future events .

ELIGIBILITY:
Inclusion Criteria:

* -Healthy subjects without any past or present psychiatric or neurological disorders

Exclusion Criteria:

* History of brain injury
* Psychiatric or Neurological Disorder
* Contraindications for MRI
* Regular use of psychotropic substances (medication, drugs)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-16 (Actual); Primary Completion 2026-06-10 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Neural activity of the medial prefrontal cortex (mPFC) based on blood oxygen level-dependent (BOLD) signal | 1 hour
  Training-induced changes in mPFC activity will be assessed by analyzing BOLD-level activation of the mPFC

SECONDARY OUTCOMES:
Training-related changes in anticipated anxiety | 1 hour
  Participants will be required to rate the anticipated anxiety of future events using a Likert Scale ranging from 1 to 9 (1 = not at all anxious) and 9 = very anxious).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Electronic Science and Technology of China(UESTC), Chengdu, Sichuan 611731, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No
Corresponding individual level data will be made available upon request.